CLINICAL TRIAL: NCT02621762
Title: Pilot Study to Investigate the Effects of Increased Dialysate Magnesium and Dialysate Bicarbonate on the Calcification Propensity of Serum
Acronym: BicMag
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 293_15
Record Dates: First submitted 2015-11-26; First posted 2015-12-03 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: End Stage Renal Failure on Dialysis; Vascular Calcification
MeSH Terms: conditions — Vascular Calcification

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mg first (Experimental): Receives MgCl2 first, MgCl2 and Bicarbonate in second phase
  Interventions: Device: Magnesium; Device: Bicarbonate
- Bicarbonate first (Experimental): Receives Bicarbonate first, MgCl2 and Bicarbonate in second phase
  Interventions: Device: Magnesium; Device: Bicarbonate

INTERVENTIONS:
Device: Magnesium — Magnesium in dialysate increased
Device: Bicarbonate — Bicarbonate in dialysate increased

SUMMARY:
The study aims to determine the effect size of magnesium and bicarbonate supplementation as a basis for future randomized controlled trials aiming at the T50-guided improvement of hard clinical endpoints in dialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female hemodialysis patients ≥ 18 years of age
* Negative pregnancy test of female patients in child-bearing age
* The patients have to be able to understand the character and the individual impact of the clinical study and they have to give written informed consent to participate in the study
* Start of chronic hemodialysis treatment ≥ 3 months ago
* HCO3- in venous plasma ≤23 mmol/L before the start of the last dialysis of the week
* Magnesium in venous plasma ≤ 1.45 mmol/L before the start of the first dialysis of the week
* T50 ≥ 200 minutes.

Exclusion Criteria:

* Pregnant or lactating subjects. A blood pregnancy test will be performed at the screening visit in female patients of childbearing age.
* History of alcohol abuse, illicit drug use, significant mental illness, physical dependence to any opioid, or any history of drug abuse or addiction within 12 months of study enrolment

Ages: 18 Years to 111 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-12; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Effect of treatment on serum calcification propensity, measured by T50 | 7 weeks
  T50: Transformation time of primary calciprotein particles to secondary calciprotein particles (Pasch et al, 2012)

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events | 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dominik Uehlinger, Prof Dr.med., Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (1):
- University Hospital Bern Inselspital, Bern, Canton of Bern, Switzerland

REFERENCES:
- [Background] Pasch A, Farese S, Graber S, Wald J, Richtering W, Floege J, Jahnen-Dechent W. Nanoparticle-based test measures overall propensity for calcification in serum. J Am Soc Nephrol. 2012 Oct;23(10):1744-52. doi: 10.1681/ASN.2012030240. Epub 2012 Sep 6. PMID 22956818